CLINICAL TRIAL: NCT03168009
Title: The Role of Alternatively Activated Brown Fat in Bariatric Surgery-mediated Metabolic Improvements
Brief Title: Brown Fat Activity and Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Florian Kiefer, Associate Professor of Medicine, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1071/2017
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Obesity
Keywords: BAT; Bariatric Surgery; Energy Metabolism
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bariatric Surgery (Experimental): Patients will undergo either Omega Loop Gastric Bypass or Sleeve Gastrectomy. The decision which type of surgery will be performed, will by made by the surgeon and the patient based on clinical considerations and the patient's wishes.
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery — Patients will undergo bariatric surgery as routinely scheduled. The type of bariatric procedure will be suggested by the surgeon based on clinical considerations.

SUMMARY:
The mechanisms of bariatric surgery-induced weight loss go beyond reductions in calorie intake and may involve several other pathways. Recently, brown adipose tissue (BAT) has been added as another potential player. Activation of BAT results in enhanced energy expenditure and promotes weight loss. Here, the investigators will study the effects of bariatric surgery on BAT function by PET/CT studies and molecular analyses of adipose biopsies. The investigators will explore different pathways that may affect BAT activation in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 50 years
* Body mass index (BMI) 35 - 55kg/m2

Exclusion Criteria:

* Endocrine disease (except hyperlipidemia and substituted hypothyroidism or type 2 diabetes with fasting glucose concentrations <120mg/dl), kidney disease, inflammatory bowel disease, autoimmune or rheumatologic diseases that require immunosuppressive treatment, active oncologic disease, heart failure.
* Medication for any of the above mentioned conditions.
* Antibiotic treatment in the past three months
* Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in BAT activity after bariatric surgery | 4 years
  The primary outcome of this study is to determine whether Omega Loop Gastric Bypass and Sleeve Gastrectomy result in increased BAT activity

SECONDARY OUTCOMES:
Bariatric surgery-induced changes in gut microbiota, bile acid composition and other circulating factors | 4 years
  Any pre-versus postsurgical changes of the gut microbiota or bile acid composition or other circulating factors will be evaluated.
Association between changes in BAT activity, transcriptional BAT markers and alterations in the gut microbiota profile or bile acid composition | 4 years
  Linear regression analyses will be performed to determine any association between BAT activity or molecular signature and changes in the gut microbiota or bile acids

CONTACTS AND LOCATIONS:
Overall Officials: Florian Kiefer, MD,PHD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Herz CT, Kulterer OC, Prager M, Marculescu R, Prager G, Kautzky-Willer A, Hacker M, Trajanoski S, Kofeler HC, Galle B, Haug AR, Berry D, Kiefer FW. Bariatric surgery promotes recruitment of brown fat linked to alterations in the gut microbiota. Eur J Endocrinol. 2025 Apr 30;192(5):603-611. doi: 10.1093/ejendo/lvaf081. PMID 40366070